CLINICAL TRIAL: NCT02597153
Title: A Single-arm, Open, Multi-center Phase II Clinical Trial of Mitoxantrone HCL Liposome Injection in Subjects With Relapsed Cutaneous T Cell Lymphomas
Brief Title: Phase II Clinical Study of PLM60 for the Treatment of Cutaneous T Cell Lymphomas
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Just one subject enrolled in this trial during one and a half years.
Sponsor: CSPC ZhongQi Pharmaceutical Technology Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSPC-HE154/PRO/Ⅱ
Record Dates: First submitted 2015-11-03; First posted 2015-11-05 (Estimated); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Relapsed Cutaneous T Cell Lymphom

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Mitoxantrone HCL Liposome Injection (Experimental): Each treatment cycle lasts for 28 days with 20mg/m2
  Interventions: Drug: Mitoxantrone HCL Liposome Injection

INTERVENTIONS:
Drug: Mitoxantrone HCL Liposome Injection

SUMMARY:
To study efficacy and safety of Mitoxantrone HCL Liposome Injection in patients with relapsed cutaneous T cell lymphomasell

ELIGIBILITY:
Inclusion Criteria:

* The subjects are voluntary and sign the informed consent form;
* ECOG score 0 to 2;
* The expected survival time ≥3 months;
* Patients with cutaneous T-cell lymphoma confirmed by histopathology, with measurable lesions, with or without systemic lymph node involvement; clinical stage IB-IVA;
* The patients previously receive at least once of systemic therapy (including systemic electron beam irradiation or chemotherapy, stem cell transplantation) and do not achieve remission (including remission period shorter than 30 days after the treatment;
* An interval of at least four weeks after the target tumor was treated with chemotherapy, radiotherapy, biological therapy, stem cell transplantation or other study drugs;
* Subjects at childbearing age agree to take effective contraceptive measures during the study; blood pregnancy test result is negative (except infertility due to menopause or operation);
* Laboratory tests (blood routine, liver and kidney function) meet the following requirements:

  1. ANC≥ 1.5×109/L; b) PLT ≥ 75×109/L; c) Hb ≥ 9 g/dL; d) Cr) ≤ 1.5x ULN ; e) TBIL ≤ 1.5x ULN; f) AST or ALT ≤2.5 x ULN.

Exclusion Criteria:

* Pregnant or lactating women;
* An allergic history to anthracyclines or liposome drugs;
* Disease progression or recurrence after anthracycline treatment within six months before the enrollment;"
* Patients who once used mitoxantrone injection;
* Patients who have used doxorubicin (or pirarubicin) with the total cumulative dose> 360mg/m2, or epirubicin with the total cumulative dose > 600mg/m2;
* Left ventricular ejection fraction is < 50% or < the lower limit of normal; clinically significant QT interval prolongation (>450ms in male, >470ms in female); a past history of cardiac disease caused by anthracyclines; a history of severe heart disease;
* Concomitant treatment as other anticancer drugs are needed;
* With internal organ involvement (including bone marrow, central nervous system;
* Clinically active infection that can significantly affect the clinical trial;
* Within 6 weeks after organ transplantation or major organ surgery;
* Those who are inappropriate to be enrolled as evaluated by the researchers.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2015-10 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR; complete response + partial response [CR + PR]) | Up to 6 months

SECONDARY OUTCOMES:
Duration of Response (DOR) | Time from the date at which the patient's objective status is first noted to be a CR or PR to the earliest date progression is documented (assessed up to approximately 24 months)
Time to Response (TTR) | Time from the date of registration to the date at which the patient's objective status is first noted to be a CR or PR (assessed up to approximately 24 months)
Progression-free survival (PFS) | Up to a total of 24 months after first dose or until disease progression, withdrawal from study, or death
Pruritus remission rate | Up to a total of 24 months after first dose or until disease progression, withdrawal from study, or death

CONTACTS AND LOCATIONS:
Locations (1):
- Beijing Cancer Hospital, Beijing, China